CLINICAL TRIAL: NCT05481983
Title: the Effect of Clinical Exercise Training on Foot Plantar Pressure, Subtalar Joint and Gait Patterns in Pregnancy
Brief Title: Exercise Training on Gait Pattern in Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, AYŞE KAYALI VATANSEVER, Physiotherapist, MSc., Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22-4.1T/36
Record Dates: First submitted 2022-05-03; First posted 2022-08-01 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Pregnancy
Keywords: pregnancy; physiotherapy; gait analysis; clinical exercise; plantar pressure

STUDY DESIGN:
Intervention Model Description: Randomized control, single-blind
Who Masked: Participant
Masking Description: The Randomization algorithm (Maximum Allowed % Deviation = 10%) was applied using PASS software 11.0 (NCSS LLC, Kaysville, UT) to generate a randomization list that would assign participants to two groups of 52 each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Walk exercise
  Interventions: Other: Walk exercise
- study group (Active Comparator): One-on-one clinical exercise training
  Interventions: Other: One-on-one clinical exercise training

INTERVENTIONS:
Other: Walk exercise — The control group will be recommended to walk 5 days a week, 30-45 minutes (min.) (at least 150 minutes of physical activity per week), as recommended by ACOG for pregnant women. Exercise intensity will be given as 4-6 units for moderate-intensity exercise according to the Modified Perceived Difficulty Level (RPE).
  Arms: control group
Other: One-on-one clinical exercise training — One-on-one clinical exercise training will be given by a specialist physiotherapist who has received special training in antenatal exercise. The program is designed to be 2 days a week for 8 weeks.
  Arms: study group

SUMMARY:
The research will be conducted with healthy pregnant women who applied to the Ege University Gynecology and Obstetrics Department Polyclinic, and were referred to the Sports Medicine Department.The study will consist of two groups as the control group and the exercise group.Voluntary pregnant women who are not found to be inconvenient to do moderate-intensity exercise by the doctor will participate in the study.The study was planned as a randomized controlled and single-blind study.The participant's demographic information, obstetric assessment, physical activity level, fall history and pain assessment will be recorded.Foot plantar pressure, static and dynamic balance, center of pressure (COP), subtalar joint evaluation and gait evaluation will be measured by pedobarography at Ege University Orthopedics and Traumatology Department Gait Laboratory.The control group will be offered walking as recommended by ACOG for pregnant women.Clinical exercise training will be given to pregnant women in the study group by a specialist physiotherapist.

DETAILED DESCRIPTION:
Pregnancy is a condition that includes many parameters.As the gestational week progresses and the fetus grows, changes are observed in the musculoskeletal system, hormonal system and other systems of the mother's body.Mechanical pain is observed in pregnant women with the expansion of the pelvis and the increase in the load on the lower extremities.The American Society of Obstetrics and Gynecology (ACOG) recommends physical activity and moderate-intensity exercises for a healthy pregnancy and delivery in pregnant women.Foot plantar pressure measurement is accepted in the literature as an objective measurement method in lower extremity biomechanical pain, static and dynamic balance.Evaluations will be made on day 0 and the day corresponding to the end of the 8th week.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-40
* No risk of pregnancy-related complications
* Between 12th and 24th weeks of pregnancy

Exclusion Criteria:

* History of lower extremity, pelvis or spine surgery
* Pain in the lower extremity, pelvis, and spine that persists for more than 6 months
* Any developmental delay related to the fetus

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-12-28 (Estimated)

PRIMARY OUTCOMES:
Foot plantar pressure | 8 weeks
  A change in gait pattern will be observed with pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: SEÇKİN ŞENIŞIK, Doktor, Study Director — Ege University
Locations (1):
- Ege University Department of Sports Medicine, Izmir, Bornova, Turkey (Türkiye)